CLINICAL TRIAL: NCT00005725
Title: Low Literacy CVD Diet Education for Blacks
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4934; R01HL046778 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To develop and demonstrate the efficacy of a set of original, cardiovascular (CVD) nutrition education materials designed to reduce intake of sodium (Na) fat, and cholesterol and which would be appropriate for urban Black adults with 5th to 8th grade reading levels.

DETAILED DESCRIPTION:
BACKGROUND:

The study was part of an NHLBI initiative on "CVD Nutrition Education for Low Literacy Skills". The initiative originated within the Prevention and Demonstration Branch of the DECA, was approved by the September 1988 National Heart, Lung, and Blood Advisory Council, and released in July 1990.

DESIGN NARRATIVE:

Materials were designed to accomplish the objectives of conventional nutrition education/behavior change programs, but avoiding the usual dependency of traditional programs on strategies that required a high level of reading and arithmetic. Guiding principles were: the need to identify the food related conceptual, cultural, and social frameworks of members of the target audience; and develop a program that built upon already-developed, alternative communication and coping skills. The core of the system was a) a protocol for office-based patient assessment and follow up, b) an educational/motivational videotape viewed in the clinical setting, c) scripts and supporting materials for a 4-week minicourse led by a clinic staff member or volunteer, and d) a package of audiocassettes and supporting printed materials to facilitate self-directed learning over an extended time period. Printed materials emphasized the use of cards (hence the acronym 'CARDES') that delivered single concepts about nutrition or behavior change and that permitted manipulation, selection, and reorganization of information.

CARDES was developed and evaluated in cooperation with Howard University Hospital in Washington, D.C. Using a randomized two-group design and a 12-24 month follow up, serum cholesterol and blood pressure levels of persons counseled with the CARDES program were compared with values for a control group receiving usual care. Process measures described adherence outcomes and determinants. Secondary outcomes related to CVD risk factor status were also evaluated. Prior to the evaluation, a pilot study determined the best sequence for delivering the information related to dietary change (i.e., Na first, fat/cholesterol first, or concurrent). Subsequent to the evaluation and prior to development of the final system and dissemination plan, an assessment was made of the potential utility of CARDES with other black populations with low literacy skills.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-08; Study Completion 1996-05 (Actual)

REFERENCES:
- [Background] Airhihenbuwa CO, Kumanyika S, Agurs TD, Lowe A, Saunders D, Morssink CB. Cultural aspects of African American eating patterns. Ethn Health. 1996 Sep;1(3):245-60. doi: 10.1080/13557858.1996.9961793. PMID 9395569
- [Background] TenHave TR, Van Horn B, Kumanyika S, Askov E, Matthews Y, Adams-Campbell LL. Literacy assessment in a cardiovascular nutrition education setting. Patient Educ Couns. 1997 Jun;31(2):139-50. doi: 10.1016/s0738-3991(97)01003-3. PMID 9216355